CLINICAL TRIAL: NCT04313790
Title: Assessment of the Anti-inflammatory Effect of Unfractionated Heparin Administered Either by Intravenous Infusion Versus Subcutaneous Injection in Critically Ill Septic Patients. A Randomized Controlled Trial
Brief Title: Assessment of the Anti-inflammatory Effect of Heparin Infusion Versus Subcutaneous Injection in Septic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IVSCHEP
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2020-03

CONDITIONS: Sepsis; Critical Illness
Keywords: heparin infusion; DVT prophylaxis; Anti inflammatory
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin Infusion (Experimental): heparin infusion 500unit \hour
  Interventions: Drug: Heparin Infusion
- Subcutaneus Heparin (Other): subcutaneous heparin 5000unit \ 8 hours
  Interventions: Other: subcutaneous heparin

INTERVENTIONS:
Drug: Heparin Infusion — 500 unit heparin infusion \ hour for DVT prophylaxis experimental group (n=20)
  Other Names: new regimen
  Arms: Heparin Infusion
Other: subcutaneous heparin — 5000 unit subcutaneous heparin /8 hours control group n=(20)
  Other Names: conventional regimen
  Arms: Subcutaneus Heparin

SUMMARY:
Venous thromboembolism (VTE), including pulmonary embolism (PE) and deep venous thrombosis (DVT), is a common and severe complication of critical illness. Critically ill patients are at high risk of VTE because they combine both general risk factors together with specific ICU risk factors of VTE. Vasopressor administration was found to be an independent risk factor for DVT. certainly explained by reduced absorption of subcutaneous heparin linked to the vasoconstriction of peripheral blood vessels. For critically ill patients, due to the altered pharmacokinetics behavior of unfractionated heparin, continuous intravenous infusion of the low doses of unfractionated heparin has been proposed. Standard prophylaxis with subcutaneous (SC) heparin is less efficient in patients requiring vasopressors. Sepsis is a systemic inflammatory response due to an infection. Both inflammatory mediators and coagulation are involved in sepsis. the release of inflammatory mediators such as interleukins and tumor necrosis factor causes damage to the endothelium and activation of coagulation which promotes the inflammatory process. Unfractionated heparin is the most negatively charged biological molecule known, heparin has a strong ability to interfere with the functioning of positively charged molecules. Due to the difference in charges, heparin has been documented to interact with over 100 proteins.57 Interleukins, cytokines, and receptors located on endothelial cells, which are involved in the acute phase response, are positively charged and thus are a reasonable target for the modulating effects of heparin. Heparin has strong anti-inflammatory effects with many possible mechanisms, including binding to cell-surface glycosaminoglycans, preventing leukocyte migration, direct binding to chemokines and cytokines, and inhibition of intracellular NF-kB.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from the Ethics Committee of the Faculty of Pharmacy, Damanhour University.
2. All participants or their next kin should agree to participate in this clinical study and will provide informed consent.
3. 40 participants who are critically ill with sepsis.
4. The 40 participants will be randomly assigned into 2 groups:

   * Standard care group: will be treated with subcutaneous heparin 5000 units three times daily for DVT prophylaxis.
   * Experimental group: will be treated with heparin infusion 5000 unit\hour for DVT prophylaxis
5. All patients will be subjected directly at the time of enrollment to the following:

   * Full patient history and clinical examination.
   * complete blood picture, liver function tests, and renal function tests.
   * The initial cause of ICU admission and define the origin of the present infection.
   * Complete cultures obtained urine, blood, and sputum.
   * Coagulation profile (prothrombin time, prothrombin activity, international normalization ratio (INR), clotting time, and activated partial thromboplastin time).
   * Arterial blood gases analysis (including hypoxic index).
   * The severity of disease assessment using Acute Physiology and Chronic Health Evaluation version II (APACHE II) score.
   * Organ failure assessment using Organ Failure Assessment (SOFA) score and quick (SOFA) score.
   * Kidney assessment using Kidney Disease Improving Global Outcomes (KDIGO) criteria.
   * Liver disease assessment using Child-Pugh Score.
   * Chest radiography, electrocardiography, and transthoracic echocardiography.
   * Vital signs (systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate temperature, blood sugar level, and urine output).
6. All patients will be monitored for the incidence of DVT, minor and major bleeding during their intensive care unit stay (ICU).
7. Coagulation profile, serum lactate, serum electrolytes, hypoxic index,14-day mortality, and the following pro-inflammatory biomarkers will be measured at the start and at days 1,2, and 7 of the study.

   i. CRP ii. Heparin-binding protein (HBP) iii. Plasminogen activator inhibitor (PAI).
8. Patient demographic data will be recorded with respect to sex. age, weight, disease, and medication history.
9. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
10. Results, conclusion, discussion, and recommendations will be given.
11. A p-value of less than 0.05 will be considered statistically significant.
12. The study data were evaluated using IBM SPSS software (statistical product and service solution version 26.0)

ELIGIBILITY:
Inclusion Criteria:

* Adults Patients aged 18 years old or greatecritically ill patients aged 18-65 years diagnosed with sepsis/septic shock or developed sepsis/septic shock during their ICU length of stay were enrolled.

Exclusion Criteria:

-Thrombocytopenia, Intracerebral hemorrhage at the time of sepsis Bleeding tendency (INR ≥ 1.5 or PLT < 50 x 109/L,) Medical condition requiring therapeutic anticoagulation Age < 18 years Previous history of Heparin Induced Thrombocytopenia (HIT).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Dynamic changes of HBP | day one, two, and seven
  Measuring the differences of HBP dynamic changes between the two study groups
Dynamic changes of PAL-1 | day one, two, and seven
  Measuring the differences of PAL-1 dynamic changes between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Salahuddin, PHD, Study Director — Damanhour University; Aymen A Eltayar, MD, Study Director — Damanhour Teatching Hospital; Noha A El Bassiouny, PHD, Study Chair — Damanhour University; Amira B Kassem, PHD, Study Chair — Damanhour University; Nouran A Elsheikh, Pharm-D, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- amira Bisher kassem, Damanhūr Shubrā, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook D, Crowther M, Meade M, Rabbat C, Griffith L, Schiff D, Geerts W, Guyatt G. Deep venous thrombosis in medical-surgical critically ill patients: prevalence, incidence, and risk factors. Crit Care Med. 2005 Jul;33(7):1565-71. doi: 10.1097/01.ccm.0000171207.95319.b2. PMID 16003063
- [Background] Dorffler-Melly J, de Jonge E, Pont AC, Meijers J, Vroom MB, Buller HR, Levi M. Bioavailability of subcutaneous low-molecular-weight heparin to patients on vasopressors. Lancet. 2002 Mar 9;359(9309):849-50. doi: 10.1016/s0140-6736(02)07920-5. PMID 11897286
- [Background] Selby R, Geerts W. Prevention of venous thromboembolism: consensus, controversies, and challenges. Hematology Am Soc Hematol Educ Program. 2009:286-92. doi: 10.1182/asheducation-2009.1.286. PMID 20008212
- [Background] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Background] Jaimes F, De La Rosa G, Morales C, Fortich F, Arango C, Aguirre D, Munoz A. Unfractioned heparin for treatment of sepsis: A randomized clinical trial (The HETRASE Study). Crit Care Med. 2009 Apr;37(4):1185-96. doi: 10.1097/CCM.0b013e31819c06bc. PMID 19242322
- [Background] Wang C, Chi C, Guo L, Wang X, Guo L, Sun J, Sun B, Liu S, Chang X, Li E. Heparin therapy reduces 28-day mortality in adult severe sepsis patients: a systematic review and meta-analysis. Crit Care. 2014 Oct 16;18(5):563. doi: 10.1186/s13054-014-0563-4. PMID 25318353
- [Background] Lorente L, Martin MM, Borreguero-Leon JM, Sole-Violan J, Ferreres J, Labarta L, Diaz C, Jimenez A, Paramo JA. Sustained high plasma plasminogen activator inhibitor-1 levels are associated with severity and mortality in septic patients. Thromb Res. 2014 Jul;134(1):182-6. doi: 10.1016/j.thromres.2014.04.013. Epub 2014 Apr 29. PMID 24814968
- [Background] Elsayed E, Becker RC. The impact of heparin compounds on cellular inflammatory responses: a construct for future investigation and pharmaceutical development. J Thromb Thrombolysis. 2003 Feb;15(1):11-8. doi: 10.1023/a:1026184100030. PMID 14574071
- [Background] Li L, Pian Y, Chen S, Hao H, Zheng Y, Zhu L, Xu B, Liu K, Li M, Jiang H, Jiang Y. Phenol-soluble modulin alpha4 mediates Staphylococcus aureus-associated vascular leakage by stimulating heparin-binding protein release from neutrophils. Sci Rep. 2016 Jul 7;6:29373. doi: 10.1038/srep29373. PMID 27383625
- [Background] Chen S, Xie W, Wu K, Li P, Ren Z, Li L, Yuan Y, Zhang C, Zheng Y, Lv Q, Jiang H, Jiang Y. Suilysin Stimulates the Release of Heparin Binding Protein from Neutrophils and Increases Vascular Permeability in Mice. Front Microbiol. 2016 Aug 26;7:1338. doi: 10.3389/fmicb.2016.01338. eCollection 2016. PMID 27617009
- [Background] Tyden J, Herwald H, Hultin M, Wallden J, Johansson J. Heparin-binding protein as a biomarker of acute kidney injury in critical illness. Acta Anaesthesiol Scand. 2017 Aug;61(7):797-803. doi: 10.1111/aas.12913. Epub 2017 Jun 5. PMID 28585315
- [Background] Fisher J, Russell JA, Bentzer P, Parsons D, Secchia S, Morgelin M, Walley KR, Boyd JH, Linder A. Heparin-Binding Protein (HBP): A Causative Marker and Potential Target for Heparin Treatment of Human Sepsis-Induced Acute Kidney Injury. Shock. 2017 Sep;48(3):313-320. doi: 10.1097/SHK.0000000000000862. PMID 28319494
- [Background] Lin Q, Shen J, Shen L, Zhang Z, Fu F. Increased plasma levels of heparin-binding protein in patients with acute respiratory distress syndrome. Crit Care. 2013 Jul 24;17(4):R155. doi: 10.1186/cc12834. PMID 23883488